CLINICAL TRIAL: NCT06995092
Title: Rhythmic Auditory Stimulation as Pre-Gait Training for Improving Balance and Weight Shifting in Rehabilitation Patients: A Feasibility Randomized Controlled Trial
Brief Title: Rhythmic Auditory Stimulation as Pre-Gait Training for Improving Balance and Weight Shifting in Rehabilitation Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pre-Gait Training
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Acute; Gait, Spastic; Attention Impaired
Keywords: Music therapy; randomised controlled trial; rehabilitation; stroke; cognition; attention
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant - Randomised by Principal Investigator Care Provider - Music Therapist Investigator - Rehabilitation Specialist Outcome Assessor - Neuropsychologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Patient will receive a 15-minute RAS session immediately before patient standard physiotherapy session. The RAS session will consist of metronome beats matched to your walking cadence. After completing the RAS sessions, patient will continue with the standard rehabilitation program as usual.
  Interventions: Other: Music therapy
- Control group (Placebo Comparator): Patient will receive the standard physiotherapy program without the RAS pre-gait training. Therapy will include sessions aimed at improving balance and gait, conducted for 15 minutes during each session. Assessments will be conducted at baseline, after completing the therapy, and during two follow-up evaluations. stroke period focuses on restoring cognitive abilities such as attention, memory, executive functions, and communication.
  Interventions: Other: Standard physiotherapy program

INTERVENTIONS:
Other: Music therapy — Patient will receive a 15-minute RAS session immediately before patient standard physiotherapy session. The RAS session will consist of metronome beats matched to your walking cadence. After completing the RAS sessions, patient will continue with the standard rehabilitation program as usual.
  Arms: Intervention group
Other: Standard physiotherapy program — Patient will receive the standard physiotherapy program without the RAS pre-gait training. Therapy will include sessions aimed at improving balance and gait, conducted for 15 minutes during each session. Assessments will be conducted at baseline, after completing the therapy, and during two follow-up evaluations.
  Arms: Control group

SUMMARY:
The purpose of this study is to explore whether Rhythmic Auditory Stimulation (RAS) as pre-gait training can help improve balance, weight-shifting abilities, and overall gait performance in stroke patients undergoing rehabilitation.

This is a feasibility study, designed to evaluate the practicality of incorporating RAS into stroke rehabilitation programs. It aims to assess how well patients can participate in and adhere to this intervention, as well as how seamlessly it integrates with standard physiotherapy treatments typically provided to stroke patients. By examining these factors, the investigators aim to identify the resources, staff training, and planning required to implement RAS as a regular component of stroke rehabilitation in the future.

The study will also help estimate the effects of RAS on balance and gait outcomes, providing preliminary data to design a larger, more comprehensive study in the future.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability worldwide, often resulting in impairments such as balance deficits and gait abnormalities, which significantly impact patients' quality of life and independence in daily functioning. Rehabilitation for individuals with gait impairments typically involves physiotherapy aimed at improving balance and weight shifting. Rhythmic Auditory Stimulation (RAS) is an evidence-based therapeutic technique that uses rhythmic cues to enhance motor control and coordination. Preliminary studies suggest that RAS can improve gait performance, but its potential as a pre-gait training intervention prior to physiotherapy sessions has not been extensively explored.

Despite a concerted effort to promote the use of music therapy in Malaysia over the last decade, structured approaches integrating RAS into local rehabilitation programs remain lacking. This contrasts with neighboring countries such as Singapore, where music therapy has gained traction as a formal therapeutic modality.

This study proposes to investigate the feasibility and potential benefits of incorporating RAS into pre-gait training for rehabilitation patients. If successful, this approach could support the integration of RAS into clinical neurorehabilitation settings, providing a scalable and accessible solution to improve balance and weight-shifting abilities, ultimately enhancing the overall effectiveness of gait-focused physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gait impairments
* Referred to physiotherapy for rehabilitation
* Ability to provide informed consent
* Understands Bahasa Melayu or English with basic communication abilities to follow instructions during therapy sessions

Exclusion Criteria:

* Severe cognitive impairments
* Severe auditory impairments
* Severe or unstable medical conditions (e.g., uncontrolled hypertension or diabetes).
* Medications that significantly impair cognition or motor function (e.g., high-dose sedatives).
* History of neurological diseases other than stroke (eg, Parkinson's disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 3 Months
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. Cut-off scores for the elderly were reported by Berg et al 1992 as follows :
  A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. A score of ≤49 indicates a risk of falls in individuals with stroke .

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suh JH, Han SJ, Jeon SY, Kim HJ, Lee JE, Yoon TS, Chong HJ. Effect of rhythmic auditory stimulation on gait and balance in hemiplegic stroke patients. NeuroRehabilitation. 2014;34(1):193-9. doi: 10.3233/NRE-131008. PMID 24284453
- [Background] Gonzalez-Hoelling S, Bertran-Noguer C, Reig-Garcia G, Suner-Soler R. Effects of a Music-Based Rhythmic Auditory Stimulation on Gait and Balance in Subacute Stroke. Int J Environ Res Public Health. 2021 Feb 19;18(4):2032. doi: 10.3390/ijerph18042032. PMID 33669715
- [Background] Hayden R, Clair AA, Johnson G, Otto D. The effect of rhythmic auditory stimulation (RAS) on physical therapy outcomes for patients in gait training following stroke: a feasibility study. Int J Neurosci. 2009;119(12):2183-95. doi: 10.3109/00207450903152609. PMID 19916847
- [Background] Mainka S, Wissel J, Voller H, Evers S. The Use of Rhythmic Auditory Stimulation to Optimize Treadmill Training for Stroke Patients: A Randomized Controlled Trial. Front Neurol. 2018 Sep 14;9:755. doi: 10.3389/fneur.2018.00755. eCollection 2018. PMID 30271375
- [Background] Yoo GE, Kim SJ. Rhythmic Auditory Cueing in Motor Rehabilitation for Stroke Patients: Systematic Review and Meta-Analysis. J Music Ther. 2016 Summer;53(2):149-77. doi: 10.1093/jmt/thw003. Epub 2016 Apr 15. PMID 27084833